CLINICAL TRIAL: NCT01642745
Title: Mannitol and Methacholine Responsiveness: Effects of Deep Inhalations
Brief Title: Mannitol (Aridol) and Methacholine (Provocholine) Responsiveness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, College of Medicine, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: IIS-A-522
Record Dates: First submitted 2012-01-17; First posted 2012-07-17 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Methacholine Chloride; Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Methacholine (Provocholine) with deep inhalation (Experimental)
  Interventions: Drug: Methacholine (Provocholine)
- Mannitol (Aridol) (Experimental)
  Interventions: Drug: Mannitol (Aridol)
- Methacholine (Provocholine) tidal breathing (Active Comparator)
  Interventions: Drug: Methacholine (Provocholine)

INTERVENTIONS:
Drug: Methacholine (Provocholine) — two minutes of aerosol inhalation of concentrations of methacholine ranging from 0.03 - 256mg/mL
  Arms: Methacholine (Provocholine) with deep inhalation
Drug: Mannitol (Aridol) — single deep inhalation of dry powder per dose doses range from 0mg - 160mg (cumulative dose range 0mg-635mg).
  Arms: Mannitol (Aridol)
Drug: Methacholine (Provocholine) — two minutes of aerosol inhalation of concentrations of methacholine ranging from 0.03 - 256mg/mL every 20 seconds a deep inhalation is performed
  Arms: Methacholine (Provocholine) tidal breathing

SUMMARY:
The study will compare the airway responses to two bronchoconstricting agents, mannitol and methacholine.

ELIGIBILITY:
Inclusion Criteria:

* stable controlled asthma

Exclusion Criteria:

* pregnancy
* use of asthma therapies other than bronchodilator therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Airway responsiveness (PC20) to methacholine delivered over two minutes of tidal breathing | Visit 1 (Day 1)
  The two minute tidal breathing PC20 with be captured once at visit 1.
airway responsiveness (PD15) to inhaled mannitol | Visit 2 = up to 13 days
  The PD15 to mannitol will be captured once at either visit 2 or visit 3.
Airway responsiveness (PC20) to deep inhalation methacholine | Visit 3 = up to 14 days
  The PC20 to methacholine (deep inhalation) will be captured once at either visit 2 or visit 3.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis BE, Stewart SL, Martin AL, Cockcroft DW. Low levels of fractional exhaled nitric oxide and deep inhalation bronchoprotection are associated with mannitol non-responsiveness in asthma. Respir Med. 2014 Jun;108(6):859-64. doi: 10.1016/j.rmed.2014.03.005. Epub 2014 Mar 20. PMID 24702886